CLINICAL TRIAL: NCT00416936
Title: Bacterial Contamination of Anaesthetists' Hands by Personal Mobile Phones Used in the Operating Theatre
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Other Study IDs: AB_12_12_2006
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Environmental Microbiology; Equipment Contamination; Personnel, Hospital

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The use of mobile phones in the operating room (OR) has become widespread, because of the lack of reports on serious problems. Since mobile phones are used in close body contact and since, as for most non-medical electronic equipment, there are no cleaning guidelines that meet hospital standards, the hygiene risk involved in using mobile phones in the OR has not yet been determined.

ELIGIBILITY:
Inclusion Criteria:

* Anaesthetist working in the OR

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2007-01; Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf Benzer, MD, Principal Investigator — Medical University Innsbruck; Arnulf Benzer, MD, Study Director — Medical University Innsbruck
Locations (1):
- University Hospital Innsbruck, Innsbruck, Austria

REFERENCES:
- [Background] Klein AA, Djaiani GN. Mobile phones in the hospital--past, present and future. Anaesthesia. 2003 Apr;58(4):353-7. doi: 10.1046/j.1365-2044.2003.03079.x. PMID 12648117
- [Background] Soto RG, Chu LF, Goldman JM, Rampil IJ, Ruskin KJ. Communication in critical care environments: mobile telephones improve patient care. Anesth Analg. 2006 Feb;102(2):535-41. doi: 10.1213/01.ane.0000194506.79408.79. PMID 16428557
- [Background] Smith MA, Mathewson JJ, Ulert IA, Scerpella EG, Ericsson CD. Contaminated stethoscopes revisited. Arch Intern Med. 1996 Jan 8;156(1):82-4. PMID 8526701